CLINICAL TRIAL: NCT04923009
Title: Simplified Pulmonary Vein Isolation Using singLe Catheter and IntraCardiac Echocardiography: The Simple-ICE Study
Brief Title: Simplified Pulmonary Vein Isolation Using singLe Catheter and IntraCardiac Echocardiography
Acronym: Simple-ICE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, Professor, Centre of Postgraduate Medical Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMKP nr 15/2021
Record Dates: First submitted 2021-05-27; First posted 2021-06-11 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; intracardiac echocardiography
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Consecutive patients prospectively included in one of the two study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple-ICE group (Experimental): Patients undergoing ablation using only ICE visualization and ablation catheter
  Interventions: Procedure: ICE visualization and map construction
- Standard mapping catheter without ICE (Active Comparator): Patients undergoing ablation using standard approach including diagnostic and mapping electrodes as well as ablation electrode
  Interventions: Procedure: ICE visualization and map construction

INTERVENTIONS:
Procedure: ICE visualization and map construction — Radio-frequency ablation of atrial fibrillation
  Other Names: RF ablation

SUMMARY:
Ablation for paroxysmal atrial fibrillation (PAF) by means of pulmonary vein isolation (PVI) is the principal method for the treatment of PAF. Usually, PVI is confirmed by recording PV potentials (PVP) from the circular catheter placed at the ostium of PV. However, newer and faster methods became avialable. The only currently available technique which can visualize LA anatomy on-line, is intracardiac echocardiography (ICE). It seems that ICE could replace all other techniques used for LA imaging. Also, there may be no need for introducing diagnostic catheters and only ablation catheter and single transseptal puncture will do.

Hypothesis. Simplified ICE-based ablation is faster and with shorter fluoroscopy time than standard ablation without compromising safety and efficacy and with no significant increase in costs.

Aim. To compare procedural data, costs, safety and efficacy of simplified ICE-based ablation versus standard RF ablation for AF.

Methods. This is prospective, controlled trial. Three centers will be included: center 1 where simplified ICE-based procedure is performed and centers 2 and 3 where standard approach is used. Patients with PAF will be allocated to two approaches: (1) standard (n=45) arm undergoing multi-electrode RF ablation in centers 2 and 3 and (2) the simple-ICE group (n=45) undergoing RF ablation in center 1 using ablation catheter and ICE catheter only.

Ablation procedure will be performed using electro-anatomical system according to the CLOSE protocol. In the simple-ICE group PVI is confirmed by lack of LA capture during pacing from or up to 5 mm inside the ablation line. In the standard group both pacing from ablation line and signals from the circular diagnostic electrode will be used to confirm PVI.

A one year follow-up is planned including three visits in cardiology clinics with 4-7 day Holter ECG 3, 6 and 12 months after the procedure.

Assessed outcomes include duration of procedure, duration and dose of radiation, one-year procedural efficacy, peri- and post-procedural complications and cost-efficacy

DETAILED DESCRIPTION:
I. Introduction. Ablation for paroxysmal atrial fibrillation (PAF) by means of pulmonary vein isolation (PVI) is the principal method for the treatment of PAF. In the majority of centers PVI is confirmed by recording PV potentials (PVP) from the circular catheter placed at the ostium of PV. However, this method of confirming PVI by demonstrating conduction block has been developed several years ago when techniques and operator skills in creating continuous and transmural radio-frequency (RF) lesions around PV was far from optimal. Nowadays, technical progress led to significant improvement in the quality of RF lesions thanks to the advent of ablation electrodes with contact force (CF) measurement and computation of ablation index which includes stability of electrode, impedance, CF and temperature measurements. In addition, implementation of so-called CLOSE protocol and paying attention to the contiguity of RF lesions further improved the outcome of ablation. Therefore, it may be speculated that the time has come to give up using circular electrode to confirm PVI, especially that another technique to confirm PVI has been available for a long time. This technique consists of pacing from ablation electrode from the line of RF applications or slightly inside this line to confirm lack of impulse conduction from PV to the left atrium (LA). In addition, lack of PV signals from the tip of ablation electrode further confirms PVI.

Another progress in AF ablation consists of the expanding usage of electro-anatomical systems (EAM) and reconstructing LA chamber which enables performing procedure with minimal fluoroscopy. In recent years, the usual approach consisted of reconstructing LA chamber using fast electro-anatomical (FAM) technique by means of dedicated circular diagnostic electrode or, more time consuming, ablation electrode [6]. Another approach consisted of pre-procedural LA imaging using computed tomography or cardiac magnetic resonance and merging this image with the electro-anatomical map. In addition, rotational angiography for LA visualization has been used. However, all these methods have several limitations and drawbacks such as radiation exposure, additional cost and creation of LA anatomy before rather than during the ablation procedure which may not be very accurate.

The only currently available technique which can visualize LA anatomy on-line, is intracardiac echocardiography (ICE). The CartoSound software provides fast and adequate delineation of the LA chamber. It has been shown that ICE-based LA reconstruction may slightly underestimate chamber dimensions whereas FAM overestimates LA size. Also, ICE images acquired directly from the LA may improve procedural accuracy. There is no doubt that training and experience in using ICE for LA reconstruction are essential for achieving good quality LA maps. Thus, it seems that ICE could replace all above mentioned techniques used for LA imaging.

Additionally, ICE has been used during AF ablation for (1) performing safe and adequately directed transseptal puncture, (2) assessment of electrode contact with cardiac tissue, (3) choosing right spot for RF applications and (4) early detection of complications. Therefore, it is very tempting to use ICE also for creating LA anatomy as this tool has already been used during ablation procedures in many centers. Such an approach might reduce costs associated with the usage of other imaging tools and possibly shorten procedural duration. In addition, ICE can be effectively used for the LA appendage (LAA) assessment for the presence of clots and, therefore, the usage of transesophageal echocardiography (TEE) may be abandoned, further reducing costs. The reduction in fluoroscopy time when using ICE is obvious and has been confirmed by numerous authors. Although ICE has so many advantages, it has not been routinely used in many laboratories because of the need for long training and high cost of a single-use ICE probe. However, with the reduction of costs of other equipment and procedure duration the ICE-based AF ablation may occur cost effective.

During AF ablation procedure a diagnostic catheter is usually introduced to the coronary sinus (CS). It serves for pacing and as an anatomical marker during transseptal puncture performed under fluoroscopic guidance. In many centers second diagnostic electrode is introduced to the His bundle area, also as an anatomical marker facilitating transseptal puncture. However, when using ICE, the CS and His catheters are not needed because the interatrial septum is elegantly visualized by ICE. Diagnostic catheters are also used for exclusion of other arrhythmias and for urgent pacing if bradycardia or asystole occur during ablation, however, this can be also accomplished by pacing from ablation catheter.

Last element of AF ablation which underwent changes during recent years, is the number of transseptal punctures. Routinely, a double transseptal access has been used for many years in the majority of centers which enables keeping both ablation and circular catheter in the LA throughout the whole procedure and recording continuously progress in PVI. However, having in mind the above described progress in the quality of RF lesions around PVI it may be speculated that nowadays the use of diagnostic circular catheter may be not necessary and a single transseptal puncture will do. Even if an operator prefers for some reasons to confirm PVI using diagnostic circular catheter, second transseptal access is not mandatory because ablation electrode may be exchanged by diagnostic catheter after completing PVI using the same transseptal sheath. Single transseptal approach further decreases costs and safety of the procedure in terms of avoiding second puncture of the interatrial septum and potential thrombo-embolic risk associated with long lasting presence of the second electrode in the LA.

In summary, it may be speculated that after over 20 years of performing RF ablation for AF operator's experience and technical progress allow for simplification of the procedure, leading to further reduction in ablation duration, fluoroscopy time and costs without compromising safety and efficacy.

II. Hypothesis. Simplified ICE-based ablation is faster and with shorter fluoroscopy time than standard ablation without compromising safety and efficacy and with no significant increase in costs.

III. Aim To compare procedural data, costs, safety and efficacy of simplified ICE-based ablation versus standard RF ablation for AF.

IV. Methods. This is prospective, controlled trial. Three centers will be included: center 1 where simplified ICE-based procedure is performed and centers 2 and 3 where standard approach is used. In order to avoid inter-operator differences, all procedures are performed by the same two skilled operators and using the same ablation system.

1. Patients - consecutive subjects undergoing first ablation for PAF will be included and allocated into two groups.

   1. The standard group consists of consecutive patients from centers 2 and 3 undergoing first RF point-by-point ablation of PAF with the use of ablation electrode (Navistar SmartTouch), diagnostic circular catheter (LASSO navigational catheter or Pentaray catheter), diagnostic 10 pole CS catheter (Boston or Hagmed) and diagnostic 4-pole His catheter (Boston or Hagmed). In this group one transseptal puncture is performed using transseptal sheath (Abbott) and transseptal Brockenbrough needle (Abbott) under fluoroscopic guidance. The LA chamber and PV ostia will be reconstructed using the CARTO-3 electro-anatomical system and LASSO or Pentaray catheters. The PV ostia will be marked based on anatomy reconstructed by EAM, fluoroscopy and parameters derived from ablation electrode like impedance, tactile and contact force feedback.
   2. The simple-ICE group consists of consecutive patients undergoing first point-by-point RF ablation for PAF in center 1 using ablation catheter (Navistar SmartTouch) and ICE catheter (Acunav, ). Access to LA is achieved using the same equipment but only under ICE guidance. The LA chamber is reconstructed and PV ostia are marked using the Cartosound System. The fragments of LA which are not clearly visible in ICE will be reconstructed using the ablation catheter.
2. Ablation procedure. The RF point-by-point ablation is performed according to the CLOSE protocol with modified size of ablation dots which are reduced from 3 mm to 2 mm in order to enhance accuracy and contiguity of RF lesions. The PV are isolated in pairs (first right PV and then left PV) without delivering applications between the ipsilateral PV unless no PVI is achieved after completion the ablation line around PV. The ablation index settings are > 450 at anterior wall and > 350 at posterior wall. In the simple-ICE group PVI is confirmed by lack of LA capture during pacing from or up to 5 mm inside the ablation line. In the standard group both pacing from ablation line and signals from the circular diagnostic electrode will be used to confirm PVI. The pacing parameters are: contact force > 4 gram, pacing rate faster > 40% than sinus rate, pulse width of 10 miliAmper and pulse duration of 2 miliseconds. If conduction from PV to LA is present, additional RF applications along ablation line at these sites are performed and line between ipsilateral PV is designed until complete PV is achieved.
3. Follow-up. A one year follow-up is planned. Three visits in cardiology clinics with 4-7 day Holter ECG are scheduled 3, 6 and 12 months after the procedure. If a patient was on antiarrhythmic medication before ablation, it will be continued for three months and stopped at the 3-month visit if possible. Two definitions of ablation efficacy will be used: (i) clinical efficacy - no recurrence of symptomatic AF and (ii) ECG-based efficacy - no symptomatic AF recurrence, no AF > 30 sec during control Holter ECG monitoring or need for higher than pre-ablation doses of antiarrhythmic drug or starting new antiarrhythmic drug.
4. Outcomes. The main outcomes of the study include duration of procedure, duration and dose of radiation, one-year procedural efficacy assessed using two definitions, peri- and post-procedural complications and cost-efficacy analysis
5. Sample calculation Based on the assumption that procedure duration in the standard group is 220 minutes (mean time in centers 2 and 3 in 2020), in the ICE-based group is predicted to be shortened to 180 minutes, and that these goals will be achieved in 50% of standard group patients and 80% of the ICE-based group, the final calculated population will consist of 90 patients (45 subjects in each group). With 45 control patients and 45 ICE-group patients, there will be a 82% chance of detecting a significant difference at a two-sided 0.05 significance level. The study will last three years: two years up to recruitment of the last patient and third year to complete follow-up of the last patients.
6. Expected results:

The RF point-by-point PVI using ablation and ICE catheters only will be significantly shorter, with less fluoroscopy time and less equipment usage than standard approach. This will be achieved without compromising safety, efficacy and costs of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* first ablation for AF
* written informed consent.

Exclusion Criteria:

* previous AF ablations
* anticipated need for more complex ablation than PVI only
* lack of written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-05-24 (Estimated); Study Completion 2024-05-24 (Estimated)

PRIMARY OUTCOMES:
Duration of procedure | 100 - 240 minutes
  calculated from first skin puncture to sheaths removal

SECONDARY OUTCOMES:
Dose of radiation | up to 4 hours
  in miliGrays
Duration of radiation | up to 20 minutes
  Duration in minutes
One-year procedural efficacy | up to 366 days
  Time to first recurrence of AF after ablation
Peri- and post-procedural complications | up to 28 days
  Complications occurring during and up to 4 weeks after ablation
Cost-efficacy | two years
  Analysis of costs of used equipement in both study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
If individual data will be rquired by reviewers or other investigators (for example, for meta-analysis maiking) we will provide all details
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from May 2024
Access Criteria: after personal contact access criteria will be defined

REFERENCES:
- [Background] Taghji P, El Haddad M, Phlips T, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Evaluation of a Strategy Aiming to Enclose the Pulmonary Veins With Contiguous and Optimized Radiofrequency Lesions in Paroxysmal Atrial Fibrillation: A Pilot Study. JACC Clin Electrophysiol. 2018 Jan;4(1):99-108. doi: 10.1016/j.jacep.2017.06.023. Epub 2017 Sep 27. PMID 29600792
- [Background] Berte B, Hilfiker G, Moccetti F, Schefer T, Weberndorfer V, Cuculi F, Toggweiler S, Ruschitzka F, Kobza R. Pulmonary vein isolation using ablation index vs. CLOSE protocol with a surround flow ablation catheter. Europace. 2020 Jan 1;22(1):84-89. doi: 10.1093/europace/euz244. PMID 31518403
- [Background] Eitel C, Hindricks G, Sommer P, Gaspar T, Kircher S, Wetzel U, Dagres N, Esato M, Bollmann A, Husser D, Hilbert S, Zaker-Shahrak R, Arya A, Piorkowski C. Circumferential pulmonary vein isolation and linear left atrial ablation as a single-catheter technique to achieve bidirectional conduction block: the pace-and-ablate approach. Heart Rhythm. 2010;7(2):157-64. doi: 10.1016/j.hrthm.2009.10.003. Epub 2009 Oct 12. PMID 20036199
- [Background] Steven D, Sultan A, Reddy V, Luker J, Altenburg M, Hoffmann B, Rostock T, Servatius H, Stevenson WG, Willems S, Michaud GF. Benefit of pulmonary vein isolation guided by loss of pace capture on the ablation line: results from a prospective 2-center randomized trial. J Am Coll Cardiol. 2013 Jul 2;62(1):44-50. doi: 10.1016/j.jacc.2013.03.059. Epub 2013 May 1. PMID 23644091
- [Background] Caponi D, Corleto A, Scaglione M, Blandino A, Biasco L, Cristoforetti Y, Cerrato N, Toso E, Morello M, Gaita F. Ablation of atrial fibrillation: does the addition of three-dimensional magnetic resonance imaging of the left atrium to electroanatomic mapping improve the clinical outcome?: a randomized comparison of Carto-Merge vs. Carto-XP three-dimensional mapping ablation in patients with paroxysmal and persistent atrial fibrillation. Europace. 2010 Aug;12(8):1098-104. doi: 10.1093/europace/euq107. Epub 2010 Apr 17. PMID 20400766
- [Background] De Potter T Jr, Bardhaj G, Viggiano A, Morrice K, Geelen P. Three-dimensional Rotational Angiography as a Periprocedural Imaging Tool in Atrial Fibrillation Ablation. Arrhythm Electrophysiol Rev. 2014 Nov;3(3):173-6. doi: 10.15420/aer.2014.3.3.173. Epub 2014 Nov 29. PMID 26835087
- [Background] Singh SM, Heist EK, Donaldson DM, Collins RM, Chevalier J, Mela T, Ruskin JN, Mansour MC. Image integration using intracardiac ultrasound to guide catheter ablation of atrial fibrillation. Heart Rhythm. 2008 Nov;5(11):1548-55. doi: 10.1016/j.hrthm.2008.08.027. Epub 2008 Aug 29. PMID 18984531
- [Background] Rordorf R, Chieffo E, Savastano S, Vicentini A, Petracci B, De Regibus V, Valentini A, Klersy C, Dore R, Landolina M. Anatomical mapping for atrial fibrillation ablation: a head-to-head comparison of ultrasound-assisted reconstruction versus fast anatomical mapping. Pacing Clin Electrophysiol. 2015 Feb;38(2):187-95. doi: 10.1111/pace.12539. Epub 2014 Dec 2. PMID 25469451
- [Background] Kaseno K, Hisazaki K, Nakamura K, Ikeda E, Hasegawa K, Aoyama D, Shiomi Y, Ikeda H, Morishita T, Ishida K, Amaya N, Uzui H, Tada H. The impact of the CartoSound(R) image directly acquired from the left atrium for integration in atrial fibrillation ablation. J Interv Card Electrophysiol. 2018 Dec;53(3):301-308. doi: 10.1007/s10840-018-0368-5. Epub 2018 Apr 14. PMID 29656326
- [Background] Baran J, Stec S, Pilichowska-Paszkiet E, Zaborska B, Sikora-Frac M, Krynski T, Michalowska I, Lopatka R, Kulakowski P. Intracardiac echocardiography for detection of thrombus in the left atrial appendage: comparison with transesophageal echocardiography in patients undergoing ablation for atrial fibrillation: the Action-Ice I Study. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1074-81. doi: 10.1161/CIRCEP.113.000504. Epub 2013 Nov 15. PMID 24243787
- [Background] Brooks AG, Wilson L, Chia NH, Lau DH, Alasady M, Leong DP, Laborderie J, Roberts-Thomson KC, Young GD, Kalman JM, Sanders P. Accuracy and clinical outcomes of CT image integration with Carto-Sound compared to electro-anatomical mapping for atrial fibrillation ablation: a randomized controlled study. Int J Cardiol. 2013 Oct 3;168(3):2774-82. doi: 10.1016/j.ijcard.2013.03.130. Epub 2013 Apr 25. PMID 23623342
- [Background] Kulakowski P, Sikorska A, Piotrowski R, Krynski T, Baran J. Ablation for paroxysmal atrial fibrillation-real-life results from a middle-volume electrophysiology laboratory. J Interv Card Electrophysiol. 2021 Dec;62(3):549-556. doi: 10.1007/s10840-020-00937-1. Epub 2021 Jan 9. PMID 33423186
- [Result] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923